CLINICAL TRIAL: NCT06577402
Title: Observational Study on Energy Expenditure and Protein Metabolism Changes in Patients With Severe Brain Injury.
Status: Recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Attending Physician, Southeast University, China
Other Study IDs: 2024ZDSYLL109-P01
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Energy Metabolism and Muscle Mass Changes in Patients With Severe Brain Injury
MeSH Terms: interventions — Nutritional Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: nutritional support — nutritional support

SUMMARY:
Evaluation of early energy metabolism and muscle mass changes in patients with severe brain injury, the impact of nutritional therapy on metabolism and muscle mass, and their relationship with patient prognosis, to provide clinical research references for the implementation of individualized nutritional therapy in patients with severe brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe neurological critical illness admitted to the ICU, including moderate to severe acute cerebrovascular disease, severe acute craniocerebral injury and spinal cord injury, central nervous system bacterial infections, status epilepticus, neurosurgical patients requiring life support during the perioperative period, and other progressive severe neurological conditions.
* Age ≥ 18 years old.
* Receiving invasive mechanical ventilation.
* Willing to sign an informed consent form.

Exclusion Criteria:

* Women of childbearing age with a positive pregnancy test, pregnant, or lactating women.
* Chronic diseases with severe organ dysfunction or serious complications:

  1. Heart: New York Heart Association (NYHA) Functional Classification IV.
  2. Lung: Chronic respiratory failure requiring long-term oxygen therapy.
  3. Kidney: Chronic kidney disease stage 4 or 5; Liver: History of liver failure, hepatic encephalopathy, or hepatic coma, recent gastrointestinal bleeding due to portal hypertension, or Child-Pugh score ≥ 10.
* Cancer patients with cachexia, or with severe organ dysfunction due to obstruction, mass effect, compression, or those who have not undergone surgery due to difficulty or recent chemotherapy or immunotherapy within one month.
* Severe immunodeficiency or current use of potent immunosuppressants, agranulocytosis (N < 0.5×10^9/L), active hematologic malignancy, or HIV infection stage III; currently undergoing immunosuppressive induction therapy, such as antithymocyte globulin (ATG), antilymphocyte globulin (ALG), interleukin 2 receptor alpha chain antibody (IL-2RA), interleukin 6 receptor A antibody (IL-6RA), etc.; continuous use of glucocorticoids for more than 2 weeks, with a daily dose exceeding the equivalent of 200 mg of hydrocortisone.
* Acute gastrointestinal injury (AGI) grade IV, such as intestinal ischemia and necrosis, gastrointestinal bleeding leading to hemorrhagic shock, abdominal compartment syndrome (IAP > 20mmHg) requiring active decompression, etc.
* Implanted with life-sustaining devices such as a pacemaker.
* In a critical condition with an expected survival time of less than 24 hours.
* Receiving or requiring dialysis or renal replacement therapy within 6 hours (this time frame is considered to exclude patients who may have acute changes in renal function that could confound the study outcomes or who may be in a transient state that could resolve without the need for long-term dialysis or renal replacement therapy).
* Patients requiring or currently receiving extracorporeal membrane oxygenation (ECMO) treatment.
* Combined with severe and above burns: total body surface area of burns exceeding 30% or III-degree burns area exceeding 10%; or with a total area of less than 30%, but with a severe overall condition or in shock, combined injuries, or respiratory tract burns.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with critical neurological illness
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Basal Metabolic Rate | first 10 day

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided